CLINICAL TRIAL: NCT05876754
Title: An Open-Label Early Access Phase 3b Study of Ivosidenib in Patients With a Pretreated Locally Advanced or Metastatic Cholangiocarcinoma
Brief Title: An Early Access Study of Ivosidenib in Patients With a Pretreated Locally Advanced or Metastatic Cholangiocarcinoma
Acronym: ProvIDHe
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIM-95031-002; 2022-501463-40 (EudraCT Number)
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cholangiocarcinoma
Keywords: CCA; Pretreated locally advanced or metastatic cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — ivosidenib

STUDY DESIGN:
Masking Description: All patients, care providers, investigators, and outcomes assessors will know that each patient is taking the active study drug, ivosidenib.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ivosidenib (Experimental): Ivosidenib 500 mg, taken orally as two 250 mg tablets once daily for an unlimited amount of continuous 28-day cycles
  Interventions: Drug: Ivosidenib Oral Tablet

INTERVENTIONS:
Drug: Ivosidenib Oral Tablet — Ivosidenib 500 mg

SUMMARY:
A Phase 3b research study to consolidate the data that ivosidenib is safe and effective in adult patients with previously treated, locally advanced, or metastatic cholangiocarcinoma (CCA). All patients who meet inclusion criteria will be enrolled to receive ivosidenib tablets orally once daily for 28 day cycles, continuing as long as clinical benefit and consent for participation is maintained. There will be a minimum of 6 study visits from screening until the final follow-up, if one cycle of treatment is completed and consent is maintained through 18 months of follow-up. Each additional cycle completed will add one study visit, on the first day of each cycle.

DETAILED DESCRIPTION:
Ivosidenib is approved in the United States and in EU for the treatment of advanced or metastatic CCA; this study is being conducted to conslidate the data related to the safety, efficacy, and impact on quality of life for patients. This is an open-label, single-arm study of ivosidenib, which means that all patients meeting eligibility criteria will receive two 250 mg ivosidenib tablets, totaling 500mg of drug, to be taken orally, once daily, for 28 consecutive days, also referred to as one cycle. Additional cycles can continue as long as clinical benefit is confirmed by an investigator, and consent is maintained. There will be a screening visit, study visit on day 1 of each cycle, withdrawal visit within 42 days of stopping treatment, and a follow-up visit every 6 months for up to 18 months after stopping treatment. This results in a minimum of 6 study visits for the completion of one 28-day cycle of ivosidenib. One additional study visit will be added on day one of each additional cycle of treatment. Study visits will include an electrocardiogram (ECG), physical exam, tumor assessment, according to local practive at a given site and blood and urine analyses. If at any point ivosidenib is made available as a medical prescription at the patient's site, patients will be withdrawn from the study treatment and patients will be followed to collect data on overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonresectable or metastatic Cholangiocarcinoma (CCA), not eligible for curative-intent resection, transplantation, or ablative therapies
* Have a documented IDH1 R132C, R132L, R132G, R132H, or R132S gene-mutated disease
* Have tried at least 1 prior type of systemic therapy for CCA, and have recovered from any side effects
* Female patients of childbearing potential must have a negative blood pregnancy test prior to starting treatment and must agree to use 2 forms of contraception from the time they enroll to 1 month after their last dose of study drug
* Male patients with a female partner with childbearing potential must also agree to use 2 forms of contraception from the time they enroll to 1 month after their last dose of study drug

Exclusion Criteria:

* Received a prior IDH1 inhibitor
* Have received a transplant
* Have received systemic cancer treatment or radiotherapy within 2 weeks prior to Day 1 of Cycle 1
* Have received hepatic radiation, chemoembolization, and radiofrequency ablation within 4 weeks prior to Day 1 of Cycle 1
* Have ongoing brain metastases requiring steroids
* Have underwent major surgery within 4 weeks of Day 1 of Cycle 1 prior to C1D1
* Have an active hepatitis B (HBV) or hepatitis C (HCV) infections, known positive human immunodeficiency virus (HIV) antibody results, or acquired immunodeficiency syndrome (AIDS) related illness
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) from Day 1 of Cycle 1 through 28 days after last study treatment | Day 1 of cycle 1, Day 1 of each consecutive cycle, 28 days after last study treatment
  AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. All reported AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), using the latest version.
Number of Serious Adverse Events (SAEs) during the study treatment period (from Day 1 of Cycle 1 through the last study treatment intake or withdrawal of consent, whichever comes first). | Day 1 of cycle 1, Day 1 of each consecutive cycle, 28 + 14 days (maximum) after last study treatment, 6 months after last study treatment, 12 months after last study treatment, 18 months after last study treatment
  SAEs related to study drug will be collected irrespective of the time of onset. AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Number of QT prolongation events during electrocardiogram (ECG) assessed as Grade 2 or worse occurring from Day 1 of Cycle 1 through 28 days after last study treatment | Day 1 of cycle 1, week 2 of cycle 1, week 3 of cycle 1, Day 1 of each consecutive cycle, 28 days after last study treatment
  QT interval, using Fridericia's formula [QTcF], to average QTc interval > 480 to 500msec (Grade 2) or worse, as seen during an ECG. This is classified as an Adverse Event of Special Interest (AESI) for this study.
Change in Eastern Cooperative Oncology Group (ECOG) performance status (PS) score from baseline to worst value out of the post-baseline assessments. | Screening visit, Day 1 of cycle 1, Day 1 of each consecutive cycle, 28 + 14 days (maximum) after last study treatment
  ECOG PS scoring consists of Grade 0 - 5, with 0 being the patient is fully active and 5 being the patient is dead. Descriptive statistics of ECOG PS over time will be summarized by frequency. Shift tables may be provided for ECOG PS from baseline to worst value of post-baseline assessments.
Number of Adverse Events (AEs) leading to discontinuation or death from day 1 through 28 days after the last study treatment | Day 1 of cycle 1, Day 1 of each consecutive cycle, 28 days after last study treatment
  Total number of AEs that result in discontinuation from treatment or death. AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Total laboratory abnormalities using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 grading scale or the low/normal/high classifications based on laboratory normal ranges. | Screening visit, Day 1 of cycle 1, Day 1 of each consecutive cycle, 28 + 14 days (maximum) after last study treatment
  Listing of all laboratory hematology, coagulation, and chemistry data with values flagged as abnormal to show the corresponding NCI-CTCAE grades and the classifications relative to the laboratory normal ranges.
Change from baseline to the worst on-treatment value of laboratory abnormalities. | Screening visit, Day 1 of cycle 1, Day 1 of each consecutive cycle, 28 + 14 days (maximum) after last study treatment
  Abnormalities will be classified by using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 grading scale or the low/normal/high classifications based on laboratory normal ranges. Shift tables using NCI-CTCAE grades to compare baseline to the worst on-treatment value will be used. For laboratory tests, including hematology, coagulation, and chemistry, where NCI-CTCAE grades are not defined, shift tables using the low/normal/high [low and high] classification to compare baseline to the worst on treatment may be generated. On-treatment is considered from Day 1 of Cycle 1 through 28 days after the last dose.
Number of patients with vital sign values outside limits of the normal range at each time point. | Screening visit, Day 1 of cycle 1, Day 1 of each consecutive cycle, 28 + 14 days (maximum) after last study treatment
  Vital signs include systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature.
Mean change from baseline values to the worst on-treatment value of patients with vital signs outside limits of the normal range | Screening visit, Day 1 of cycle 1, Day 1 of each consecutive cycle, 28 + 14 days (maximum) after last study treatment
  On-treatment is considered from Day 1 of Cycle 1 through 28 days after the last dose. Vital signs include systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature.

SECONDARY OUTCOMES:
Progression-free survival (PFS) time beginning at enrollement | through 28 days after last treatment
  PFS is defined as the time from the date of enrollment to the date at which the disease escalates or progresses. It will be assessed using the Kaplan-Meier (KM) method curves and estimates. This will be based on tumor assessments conducted by the investigator according to local clinical practice.
Overall survival (OS) | through 28 days after last treatment
  OS is defined as the time from date of enrollment to the date of death due to any cause. It will be assessed using the Kaplan-Meier (KM) method curves and estimates.
Duration of response (DOR) | through 28 days after last treatment
  DOR is defined as the time from the date of response to either progression or death. It will be assessed using the Kaplan-Meier (KM) method curves and estimates. This will be based on tumor assessments conducted by the investigator according to local clinical practice.
Time to response (TTR) | through 28 days after last treatment
  TTR is defined as the time from the date of enrollment to the date of response. It will be assessed using the Kaplan-Meier (KM) method curves and estimates. This will be based on tumor assessments conducted by the investigator according to local clinical practice.
Change from baseline of Quality of life scores | through 28 days after last study treatment
  Measured by the validated European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Cholangiocarcinoma and Gallbladder Cancer Module (QLQ-BIL21). EORTC QLQ-BIL21, will be evaluated for patients with a baseline assessment and at least 1 post-baseline QLQ-BIL21 assessment that generates a score. Change from baseline for each time point, will be summarized using descriptive statistics.
Proportion of days at home or hospital for all patients | through 28 days after last treatment
Change from baseline of health economic measures, as assessed by the 5-level EuroQol 5-dimensional questionnaire (EQ-5D-5). | through 28 days after last treatment
  Health economic measures, as assessed by the EQ-5D-5L, will be evaluated for patients with a baseline assessment and at least 1 post-baseline EQ-5D-5L assessment that generate a score. Change from baseline scores for each time point will be quantified with descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (78):
- Armenia (2):
  - Erebouni MC, Yerevan
  - National Center of Oncology of Ra M, Yerevan
- Australia (5):
  - Royal brisbane & Women's Hospital, Brisbane
  - St Vincent's Hospital, Fitzroy
  - St John of God Hospital - Bendat Family Comprehensive Cancer Centre (BFCCC), Subiaco
  - Kinghorn Cancer Centre, Sydney
  - The Queen Elizabeth Hospital, Woodville
- Austria (4):
  - Medizinische Universitaet Graz, Graz
  - Ordensklinikum Linz GmbH, Linz
  - Universitaetsklinik fuer Innere Medizin III, mit Hämatologie, internistischer Onkologie, Hämostaseologie, Infektiologie, Rheumatologie und Onkologisches Zentrum, Salzburg
  - Medizinische Universitaet Wien Universitaetsklinik fuer Innere Medizin I, Vienna
- Belgium (4):
  - Universite Libre de Bruxelles ULB -, Brussels
  - Universitair Ziekenhuis Gent UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Cliniques Univ St Luc - Gastro-Enterology, Woluwe-Saint-Lambert
- Canada (5):
  - Tom Baker Cancer Center, Calgary
  - NSHA, QEII Health Sciences Centre, Halifax
  - London Regional Cancer Program, London
  - Princess Margaret Cancer Center, Toronto
  - Sunnybrook Health Sciences Centre, Toronto
- France (7):
  - Hôpital Privé Jean Mermoz, Lyon
  - Hopital de la Timone, Marseille
  - CHU Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nantes CHU de Nantes, Nantes
  - Institute Mutualiste Montsouris, Paris
  - CHU Bordeaux, Hôpital Haut-Lévêque, Pessac
  - CHU de Poitiers, Poitiers
- Germany (7):
  - Charite Universittsmedizin Berlin, Berlin
  - Universitaetsklinikum Carl-Gustav-Carus, Dresden
  - Klinik für Gastroenterologie, Hepatologie und Infektiologie Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Medizinische Fakultaet der Universitaet Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum der Universitaet Muenchen-Grosshadern, München
- Ireland (3):
  - Cork University Hospital, Cork
  - St. James Hospital, Dublin
  - St. Vincent's Private Hospital, Dublin
- Italy (11):
  - Policlinico S. Orsola-Malpighi, Bologna
  - AOU Careggi, Florence
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale San Raffaele, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - IRCCS Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Humanitas Research Hospital, Rozzano
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale Casa Sollievo della Sofferenza (CSS), San Giovanni Rotondo
  - A.O.U. Città della Salute e della Scienza di Torino, Turin
  - AOUI Verona - Ospedale Borgo Roma, Verona
- Netherlands (2):
  - Amsterdam UMC, location AMC, Amsterdam
  - Universiteit Maastricht UM - Maastricht University Medical Centre MUMC, Limburg
- Romania (5):
  - Institutul Clinic Fundeni, Bucharest
  - Regional Institute of Gastroenterology and Hepatology, Cluj-Napoca
  - Centrul de Oncologie Sfantu Necta, Craiova
  - Radiotherapy Center Cluj, Otopeni
  - Municipal Hospital Ploiesti, Ploieşti
- South Korea (5):
  - CHA Bundang Medical Center, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University, Seoul
  - Yonsei University Health System, Seoul
- Spain (10):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Universitari Vall d'Hebron/Vall Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Universitario Reina Sofa, Córdoba
  - Hospital General de Elche, Elche
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Marqués de Valdecilla, Santander
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
- United Kingdom (6):
  - University Hospitals Birmingham (UHB) NHS Foundation Trust - Queen Elizabeth Hospital Birmingham (QEHB), Birmingham
  - The Beatson Institute West of Scotland Cancer Research, Glasgow
  - Imperial College London, London
  - University College London Hospital NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle Upon Tyne Hospitals, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/